CLINICAL TRIAL: NCT00091260
Title: A Phase II Trial of the Immunomodulatory Drug CC-5013 for Patients With AL Amyloidosis
Brief Title: CC-5013 With or Without Dexamethasone in Treating Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaishali Sanchorawala (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Vaishali Sanchorawala, Principal Investigator, Boston Medical Center
Organization: Boston Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000385687; BUMC-H-23235 (Other: Boston University Medical Center IRB); CELGENE-RV-AMYL-PI-003 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Dexamethasone; dexamethasone acetate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- revlimid (Experimental): lenalidomide 15 mg/day, for 21 days with 7 days rest (28 day cycle) with or without dexamethasone 20 mg daily (10 mg BID) on Days 1-4, 9-12, and 17-20 of every other 28-day cycle.
  Interventions: Drug: dexamethasone; Drug: lenalidomide

INTERVENTIONS:
Drug: dexamethasone — dexamethasone 20 mg daily (10 mg BID) on Days 1-4, 9-12, and 17-20 of every other 28-day cycle.
  Other Names: dexamethasone acetate
Drug: lenalidomide — 15 mg/day, for 21 days with 7 days rest (28 day cycle) with or without dexamethasone
  Other Names: revlimid; CC-5013

SUMMARY:
RATIONALE: Drugs such as CC-5013 and dexamethasone may be effective in treating primary systemic amyloidosis.

PURPOSE: This phase II trial is studying CC-5013 to see how well it works with or without dexamethasone in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the tolerability of CC-5013 in patients with primary systemic (AL) amyloidosis.
* Determine the objective hematologic response rate in patients treated with this drug.
* Determine amyloid organ disease response in patients treated with this drug.

Secondary

* Determine hematologic and amyloid organ disease response in patients who do not achieve a response to CC-5013 alone and are subsequently treated with CC-5013 and dexamethasone.
* Determine the toxicity of CC-5013 in combination with dexamethasone in these patients.

OUTLINE: Patients receive oral CC-5013 once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients not achieving a hematologic response continue to receive CC-5013 as before and also receive oral dexamethasone twice daily on days 1-4, 9-12, and 17-20 of every other 28-day course for up to 6 courses of combination therapy. Patients who maintain a hematologic response after 6 courses of combination therapy may receive CC-5013 alone in the absence of disease progression or unacceptable toxicity. Patients not achieving a hematologic response after the initiation of dexamethasone are removed from the study.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 5-12.5 months.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed primary systemic (AL) amyloidosis

  * Tissue amyloid deposits or positive fat aspirate
* Meets 1 of the following criteria for AL type disease:

  * Serum or urine monoclonal protein by immunofixation electrophoresis
  * Plasmacytosis of bone marrow by monoclonal staining for kappa- or lambda-light chain isotype

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* SWOG 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood count> 3,000/mm^3
* Hemoglobin > 8 g/dL
* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 1,000/mm^3

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2 times ULN

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior thalidomide for AL amyloidosis allowed

Chemotherapy

* More than 4 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* Prior steroids for AL amyloidosis allowed

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Prior surgery allowed

Other

* Recovered from all prior therapy

Exclusion Criteria:

* No secondary or familial amyloidosis
* No multiple myeloma, defined as ≥ 30% plasma cells in bone marrow biopsy specimen OR lytic bone lesions
* No prior CC-5013

Renal

* No dialysis

Cardiovascular

* No symptomatic cardiac arrhythmia
* No oxygen-dependent restrictive cardiomyopathy

Other

* No untreated or uncontrolled infection
* No other malignancy except basal cell skin cancer or carcinoma in situ of the cervix or breast
* No other serious medical illness that would preclude study participation
* No history of hypersensitivity reaction to thalidomide
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-01; Primary Completion 2012-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Seldin, MD, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Cancer Research Center at Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lichtman EI, Seldin DC, Shelton A, Sanchorawala V. Single agent lenalidomide three times a week induces hematologic responses in AL amyloidosis patients on dialysis. Am J Hematol. 2014 Jul;89(7):706-8. doi: 10.1002/ajh.23722. Epub 2014 Apr 10. PMID 24668858

RESULTS

PARTICIPANT FLOW:
Groups:
- Revlimid: lenalidomide 15 mg/day, for 21 days with 7 days rest (28 day cycle) with or without dexamethasone 20 mg daily (10 mg twice daily) on Days 1-4, 9-12, and 17-20 of every other 28-day cycle.
  dexamethasone: dexamethasone 20 mg daily (10 mg twice daily) on Days 1-4, 9-12, and 17-20 of every other 28-day cycle.
  lenalidomide: 15 mg/day, for 21 days with 7 days rest (28 day cycle) with or without dexamethasone
Period: Overall Study
Arm/Group | Revlimid
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Revlimid
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 24
Gender [Count of Participants; unit: Participants]
  Female | 29
  Male | 53
Dialysis y/n [Count of Participants; unit: Participants]
  on dialysis | 7
  Not on dialysis | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Removed From Study Treatment Due to Toxicities
Time Frame: 1 year
Population: Number of patients who had at least one dose of CC-5013
Measure: Number; unit: participants
Arm/Group | Revlimid
Number analyzed (Participants) | 82
participants | 31

2. Primary Outcome: Number of Patients With Hematologic Response With Single-agent CC-5013
Description: Complete response = Absence of detectable monoclonal protein in serum or urine by immunofixation electrophoresis, less than 5% plasma cells on bone marrow biopsy without clonal dominance of kappa or lambda isotype, and normal serum free light chain assay.
  Partial response= For patients with detectable and quantifiable monoclonal marrow plasmacytosis= a reduction of 50% or more in plasma cells as a percentage of nucleated bone marrow cells. For patients with a detectable monoclonal peak on serum or urine protein electrophoresis= a reduction in the peak height of 50% or more.
  For patients with quantifiable urinary kappa or lambda chain concentration= a 50% reduction in daily light chain excretion in 24 hour urine.
  For patients with an elevated serum free light chain assay, a reduction of 50% or more.
Time Frame: 3 months
Population: Participants who received at least 3 cycles of single-agent CC-5013 and underwent subsequent evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid
Number analyzed (Participants) | 24
Participants | 5

3. Secondary Outcome: Number of Patients Who Received Both CC-5013 and Dexamethasone and Had a Hematologic Response
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Revlimid
Number analyzed (Participants) | 43
participants | 26

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Revlimid
Serious Adverse Events (participants affected / at risk) | 82/82
Other Adverse Events (participants affected / at risk) | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Revlimid (N=82)
neutropenia (Blood and lymphatic system disorders) | 15 (18)
leukopenia (Blood and lymphatic system disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
hypotension (Cardiac disorders) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
organ rejection (Cardiac disorders) | 1/1 (1) — rejection of previously transplanted heart
cardiac, other (Cardiac disorders) | 5 (5)
Fatigue (General disorders) | 18 (18)
Decreased Performance Status (General disorders) | 15 (15)
fever/infection (Infections and infestations) | 4 (6)
rash (Skin and subcutaneous tissue disorders) | 9 (10)
Nail Changes (General disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3)
dysphagia (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
infection (Infections and infestations) | 19 (19) — upper respiratory infection
increased creatinine (Renal and urinary disorders) | 6 (8)
decreased phosphate (Investigations) | 13 (13)
increased INR (Infections and infestations) | 2 (2)
muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (General disorders) | 6 (6)
pancreatitis (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
thrombosis (Vascular disorders) | 6 (6)
gout (General disorders) | 4 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid (N=82)
neutropenia (Blood and lymphatic system disorders) | 26 (32)
leukopenia (Blood and lymphatic system disorders) | 21 (26)
anemia (Blood and lymphatic system disorders) | 52 (53)
thrombocytopenia (Blood and lymphatic system disorders) | 27 (31)
hypotension (Cardiac disorders) | 7 (9)
Chest pain (Cardiac disorders) | 7 (7)
cardiac, other (Cardiac disorders) | 5 (5)
fatigue (General disorders) | 54 (61)
drowsiness (General disorders) | 11 (15)
Decreased performance status (General disorders) | 30 (30)
fever/infection (Infections and infestations) | 21 (23)
Insomnia (General disorders) | 39 (39)
Weight change (General disorders) | 16 (19)
rash (Skin and subcutaneous tissue disorders) | 29 (30)
itching (Skin and subcutaneous tissue disorders) | 22 (23)
Hot flashes (General disorders) | 4 (4)
Derm/skin other (Skin and subcutaneous tissue disorders) | 7 (7)
cushingoid (Endocrine disorders) | 4 (4)
Anorexia (Gastrointestinal disorders) | 14 (14)
early satiety (Gastrointestinal disorders) | 18 (18)
Change in appetite (Gastrointestinal disorders) | 12 (12)
constipation (Gastrointestinal disorders) | 31 (33)
diarrhea (Gastrointestinal disorders) | 30 (34)
dysphagia (Gastrointestinal disorders) | 4 (4)
dry membranes (General disorders) | 13 (13)
hemorrhoids (Gastrointestinal disorders) | 13 (13)
dyspepsia (Gastrointestinal disorders) | 17 (17)
nausea (Gastrointestinal disorders) | 24 (28)
vomiting (Gastrointestinal disorders) | 13 (15)
GI other (Gastrointestinal disorders) | 8 (8)
hemorrhage - nose (Gastrointestinal disorders) | 8 (8)
Easy bruising (Skin and subcutaneous tissue disorders) | 17 (17)
pulmonary infection (Infections and infestations) | 26 (28)
sinusitis (Infections and infestations) | 10 (10)
edema (Blood and lymphatic system disorders) | 41 (41)
hyponatremia (Investigations) | 14 (17)
hypokalemia (Investigations) | 15 (15)
increased creatinine (Investigations) | 40 (40)
hyperglycemia (Investigations) | 43 (45)
hyperbilirubinemia (Investigations) | 7 (7)
increased alkylase phosphate (Investigations) | 24 (31)
increased alanine aminotransferase test (Investigations) | 17 (17)
hypoalbuminemia (Investigations) | 33 (39)
hypocalcemia (Investigations) | 31 (31)
muscle cramps (Musculoskeletal and connective tissue disorders) | 53 (53)
numbness - extremities (Nervous system disorders) | 11 (11)
muscle weakness (Musculoskeletal and connective tissue disorders) | 16 (16)
pain - muscle (Musculoskeletal and connective tissue disorders) | 9 (9)
pain - extremities (Nervous system disorders) | 10 (10)
mood alteration (Psychiatric disorders) | 10 (10)
dizziness (General disorders) | 42 (45)
tremors (General disorders) | 6 (6)
spasms (Musculoskeletal and connective tissue disorders) | 8 (8)
tingling - extremities (Nervous system disorders) | 17 (17)
visual disturbance (Eye disorders) | 11 (11)
headache (General disorders) | 12 (12)
sore throat (Respiratory, thoracic and mediastinal disorders) | 13 (13)
cough (Respiratory, thoracic and mediastinal disorders) | 25 (25)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (28)
dysuria (Renal and urinary disorders) | 5 (5)
flu-like syndrome (General disorders) | 11 (11)
post nasal drip (Immune system disorders) | 19 (19)
elevated blood urea nitrogen blood test (Investigations) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes